CLINICAL TRIAL: NCT04700202
Title: Identifying Risk Factors for Gram-negative Resistance for HAP/VAP in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 046.PHA.2020.D
Record Dates: First submitted 2020-09-22; First posted 2021-01-07 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Ventilator-associated Pneumonia; Hospital-acquired Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective Cohort: Patients admitted to MDMC ICU from 4/1/2017 to 6/30/2020 will be identified through the electronic medical record utilizing ICD codes for HAP and VAP.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Single center, retrospective chart review. Patients admitted to MDMC ICU from 4/1/2017 to 6/30/2020 will be identified through the electronic medical record utilizing ICD codes for HAP and VAP

SUMMARY:
Single center, retrospective chart review. Patients admitted to MDMC ICU from 4/1/2017 to 6/30/2020 will be identified through the electronic medical record utilizing ICD codes for HAP and VAP.

DETAILED DESCRIPTION:
Single center, retrospective chart review. Patients admitted to MDMC ICU from 4/1/2017 to 6/30/2020 will be identified through the electronic medical record utilizing ICD codes for HAP and VAP. Patients with respiratory culture data signifying a Gram-negative organism as the cause of HAP/VAP will be analyzed as described below if study inclusion criteria is met. Minimum inhibitory concentration (MIC) data will interpreted per Clinical & Laboratory Standards Institute (CLSI) standards to determine local patterns of resistance. Multivariable logistic regression will be performed to determine risk factors for piperacillin-tazobactam, cefepime or meropenem resistant Gram-negative isolates. Project target date of completion and close-out is May 2021.

ELIGIBILITY:
Inclusion Criteria:

* ICU, Neuro critical care unit admission
* Diagnosis of HAP or VAP
* Respiratory culture positive for Gram-negative organism

Exclusion Criteria:

* ICU length of stay <48 hours prior to HAP/VAP
* Culture or MIC data unavailable
* Pregnant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to MDMC ICU from 4/1/2017 to 6/30/2020 will be identified through the electronic medical record utilizing ICD codes for HAP and VAP.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Rate of Gram-negative isolate resistance to piperacillin-tazobactam, cefepime, meropenem | April 2017 - May 2020
  Percentage

SECONDARY OUTCOMES:
Rate of susceptibility to non-beta lactam antipseudomonal agents | April 2017 - May 2020
  Percentage
in-hospital mortality | April 2017 - May 2020
  Percentage
need for mechanical ventilation | April 2017 - May 2020
  Percentage
duration of mechanical ventilation | April 2017 - May 2020
  number of days
development of septic shock | April 2017 - May 2020
  Percentage
ICU length of stay | April 2017 - May 2020
  number of days
hospital length of stay | April 2017 - May 2020
  number of days

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Crotty, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No